CLINICAL TRIAL: NCT00061711
Title: Alternative Therapies for Menopause: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: AG0003; 5R01AG017057-03 (NIH)
Record Dates: First submitted 2003-06-03; First posted 2003-06-04 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Menopause; Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — Hormone Replacement Therapy; black cohosh root extract

INTERVENTIONS:
Drug: Hormone Replacement Therapy
Drug: Cimicifuga racemosa (Black Cohosh)
Drug: Multibotanical phytoestrogen formula

SUMMARY:
This randomized, controlled trial will evaluate the efficacy and safety of three alternative approaches utilizing phytoestrogens to treat hot flashes and night sweats in peri- and post-menopausal women. The treatments were chosen because of the scientific evidence supporting a possible benefit, the availability of products with adequate quality control, and their frequency of use in naturopathic medicine. RECRUITMENT FOR THIS STUDY SHOULD END BY AUGUST 1, 2003.

DETAILED DESCRIPTION:
Over 17 million U.S. women are in the peri- and post-menopausal age range (45 - 55), and by the year 2015 nearly half of U.S. women will be post-menopausal. Of these, 25-33% will experience moderate to severe menopausal symptoms, and all will be faced with decisions related to maintaining their health through mid-life and beyond. Hormone Replacement Therapy (HRT) is the standard pharmacologic intervention for menopausal symptoms against which other therapies are measured. Concerns about breast cancer and thromboembolism risk, the need for safe alternatives for symptom relief among women in whom HRT is contraindicated, and the resistance to HRT due to its side effects fuel the search for alternatives.

The primary aim of this randomized, controlled trial is to compare the effects of three alternative treatments utilizing phytoestrogens, HRT, and placebo on the frequency and intensity of vasomotor symptoms measured by the Wiklund Menopause Symptom Checklist and daily vasomotor symptom diaries. The alternative treatments chosen for the study are a single herbal formula of black cohosh, a multibotanical formula containing black cohosh, alfalfa, boron, chasteberry, dong quai, false unicorn, licorice, oats, pomegranate, and Siberian ginseng, and soy diet counseling in addition to the multibotanical formula.

The findings of the Women's Health Initiative study published in July 2002 gave the medical and research communities new information about the long-term risk of HRT use. In response to these findings, the study design allows women to be randomized either to the 5-arm trial that includes HRT, or to be randomized only to 4 of the 5 arms: one of the three herbal groups or placebo, without the chance of being assigned to HRT.

Secondary aims are to compare the effects of three alternative treatments, HRT, and placebo on:

1. vaginal cytology (vaginal maturation index)
2. serum lipids (total cholesterol, HDL and LDL cholesterol, triglycerides)
3. bone mineral density (hip and spine dual energy x-ray absorptiometry scan)
4. glucose metabolism (insulin, fasting blood glucose)
5. clotting factors (fibrinogen, PAI-1).

Approximately 400 peri- and post-menopausal women will be recruited and randomized to one of 5 or one of 4 treatment arms for one year. Primary and secondary outcomes will be measured at baseline, 3, 6, and 12 months. Changes in outcomes will be compared between the groups taking alternative treatments and those in the HRT and placebo groups.

ELIGIBILITY:
Inclusion Criteria

1. Female, aged 45-55.
2. Peri- or post-menopausal, defined as having no menstrual periods for at least 12 months prior to study entry, or skipping at least one menstrual period in the 12 months prior to study entry. Peri- or post-menopausal status will be determined for candidates who have had the uterus removed by an assessment of blood follicle stimulating hormone (FSH). Women with an FSH level higher than 20 mlU/mL will be eligible for the study.
3. Experiencing an average of 2 or more hot flashes or night sweats per day, of which 6 or more must be of moderate or greater intensity over two weeks.
4. Normal thyroid stimulating hormone (TSH) measured prior to study entry, defined as 0.4 - 5.0 ulU/ML.
5. Proof of negative mammogram within two years prior to randomization. Subjects may provide copies of the mammogram results or a letter from their primary care provider.
6. Must provide informed consent.
7. Not at high risk for medical complications that might affect the subject's ability to complete the trial without a serious co-morbid event, based on medical history, physical examination and laboratory screening evaluation.

Exclusion Criteria

1. Mentally or legally incapacitated such that informed consent cannot be obtained.
2. Use of hormone replacement therapy or oral contraceptives within the past three months.
3. Use of alternative or complementary medicines or herbs for menopausal symptoms within the past one month.
4. History of any illness or having significant abnormalities on prestudy clinical or laboratory evaluation such that in the opinion of the investigator participating in this study might pose an unacceptable risk to the subject.
5. The subject has a medical history of any of the following contraindications to HRT: breast cancer, uterine cancer, endometrial hyperplasia, angina treated with medication, myocardial infarction, revascularization surgery, coronary angioplasty, stroke, blood clots, active chronic liver disease, or nephrotic syndrome.
6. Bone mineral density of the hip or spine more than two standard deviations below the age-specific mean.
7. bilateral oophorectomy.
8. Current use of any of the following medications: tamoxifen, raloxifene, bisphosphonates, cholesterol-lowering medications, prescription blood-thinners, or oral steroids.
9. Pregnant or planning to become pregnant.
10. Baseline blood pressure greater than 160/95 mm Hg.
11. Alergy to soybeans or soy protein.
12. Unable to swallow pills.
13. Current participation in another investigational drug trial.
14. Intention to move within the next 12 months rendering follow-up per the protocol impossible.
15. Noncompliance in the procedures involved with the screening visit or run-in trial. To be compliant, subjects must take at least 80% of the run-in medication (can miss 2-1/2 days) and complete at least 80% of the baseline symptom diaries (can miss 3 days of the hot flash and night sweats diaries, must complete all Wiklund checklists).

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 355
Dates: Start 2000-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Health Studies Research Clinic, Seattle, Washington, United States

REFERENCES:
- [Background] Newton KM, Buist DS, Keenan NL, Anderson LA, LaCroix AZ. Use of alternative therapies for menopause symptoms: results of a population-based survey. Obstet Gynecol. 2002 Jul;100(1):18-25. doi: 10.1016/s0029-7844(02)02005-7. PMID 12100799
- [Background] Phelan EA, Buist DS, Anderson LA, Newton KM, Delaney KM, LaCroix AZ. Understanding attitudes of older women toward hormone replacement therapy. Prev Med. 2001 Jan;32(1):49-56. doi: 10.1006/pmed.2000.0768. PMID 11162326
- [Background] Newton KM, LaCroix AZ, Leveille SG, Rutter C, Keenan NL, Anderson LA. Women's beliefs and decisions about hormone replacement therapy. J Womens Health. 1997 Aug;6(4):459-65. doi: 10.1089/jwh.1997.6.459. PMID 9279834
- [Background] Newton KM, LaCroix AZ, Buist DS, Keenan NL. The use of alternative and complementary medicine by women enrolled in an HMO setting. Menopause, 1998, 5:244.
- [Result] Newton KM, Reed SD, Grothaus L, Ehrlich K, Guiltinan J, Ludman E, Lacroix AZ. The Herbal Alternatives for Menopause (HALT) Study: background and study design. Maturitas. 2005 Oct 16;52(2):134-46. doi: 10.1016/j.maturitas.2005.01.007. PMID 16186076